CLINICAL TRIAL: NCT00715845
Title: Effects of Carbon Dioxide Insufflation on Cerebral Microemboli During Cardiopulmonary Bypass: A Randomised Trial Correlating Embolic Load & Neurologic Outcomes.
Brief Title: Carbon Dioxide Insufflation on Cerebral Microemboli
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: ran out of funding
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CO200
Record Dates: First submitted 2008-06-17; First posted 2008-07-15 (Estimated); Last update posted 2011-10-26 (Estimated); Status verified 2011-10

CONDITIONS: Cardiovascular Disease; Mitral Valve Repair; Cerebral Microemboli; Cognitive Decline
Keywords: cardiovascular disease; embolism; microemboli; cognitive decline; mitral valve repair; cerebral microemboli; coronary artery bypass graft; CABG; transcranial doppler; transesophageal echocardiogram; magnetic resonance imaging; carbon dioxide
MeSH Terms: conditions — Cardiovascular Diseases; Cognitive Dysfunction; Embolism | interventions — Heart-Lung Machine; Oxygenators, Membrane; Ultrasonography, Doppler, Transcranial; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- 2 (Experimental)
  Interventions: Procedure: Carbon dioxide insufflation

INTERVENTIONS:
Procedure: Carbon dioxide insufflation — For baseline evaluations, all patients will undergo a battery of neuropsychological testing after obtaining written informed consent and before cardiac surgery. A transesophageal echocardiography and a transcranial doppler will be performed for intraoperative evaluations. For post-operative evaluations, patients will undergo a diffusion-weighted magnetic resonance imaging three to seven days after surgery and have a repeat neuropsychological assessment at six to eight weeks post cardiac surgery. All patients will undergo cardiopulmonary bypass using the same equipment and technique. Patients in both groups will receive a jackson-pratt drain as a gas diffuser. The jackson-pratt drain will be placed 5 cm below the cardiothoracic wound opening adjacent to the diaphragm and if the patient is randomized to carbon dioxide, the flow will be set at 2 litre/min.
  Other Names: transeophageal echocardiogram (agilent sonos 5500); cardiopulmonary bypass circuit (sorin S3 roller pump); cardiotomy suction reservoir (dideco); membrane oxygenator (gish vision); transcranial doppler (spencer technologies PMD 100); magnetic resonance imaging (GE)

SUMMARY:
The purpose of this study is to determine if blowing carbon dioxide into the surgical field during open-heart surgery to displace retained chest cavity air from the atmosphere will decrease the number of microembolic being introduced into the heart chambers and brain.

DETAILED DESCRIPTION:
Although open-heart surgery is widely used throughout the world, from 1 to 4% of patients experience neurological impairment such as impairment of memory, language and motor skills after surgery. The cause for such cognitive impairment is thought to be air microemboli (very small bubbles of air) being introduced into the blood circulation of the brain from the heart. These air microemboli are introduced from the surgical field and/or from the heart-lung machine. During open-heart surgery, a patient's blood circulation is supported by a heart-lung machine (cardiopulmonary bypass) while the surgeon is replacing or repairing a valve or performing coronary artery bypass surgery. During valve surgery, chambers of the heart are open to room air, causing an introduction of air into the heart. Despite careful de-airing (removal of air) procedures during open-heart surgery, studies revealed that air microemboli are still formed. Past research studies have shown that carbon dioxide (CO2) filling the chest cavity by means of gravity and replacing the room air may help to decrease the amount of microemboli reaching the brain.

CO2 is 50% heavier than room air. Unlike room air, CO2 dissolves more quickly in blood and tissue (> 25 times more soluble in blood and tissue than air) whereas air contains nitrogen, which does not dissolve easily in the blood. In either case, the emboli made of air or CO2 can block the arteries of the brain causing cognitive impairment. Due to the properties of air and CO2, CO2 emboli may be tolerated much better than air emboli.

This is a single-centre, double-blind, placebo-controlled study, randomizing 100 patients undergoing elective mitral valve repair +/- coronary artery bypass grafting. Patients will be divided into 2 groups: (n=100), 50 patients will be receiving carbon dioxide insufflated and 50 patients will not. The number of microemboli will be ascertained by an intraoperative transesophageal echocardiography and transcranial doppler. Three to seven days after surgery, a magnetic resonance imaging of the brain will be done to assess for any cerebral ischemic lesions. Plus, a battery of neuropsychologic tests will be done preoperatively and 2 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* provide informed consent
* male or female who are 18 years of age or older
* elective patients to undergo mitral valve repair +/- coronary artery bypass surgery
* ability to read and write

Exclusion Criteria:

* patients with a history of stroke, TIA, carotid vascular disease
* patients with a contraindication to TEE or MRI
* patients with an active history of drug/alcohol dependence or abuse history

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-04; Primary Completion 2010-04 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Primary outcome will be the number of emboli as measured by transesophageal echocardiogram and transcranial doppler. | intraoperative

SECONDARY OUTCOMES:
Secondary outcome will be the prevalence of new ischemic lesions on diffusion weighted magnetic resonance imaging and neuropsychological impairments | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Murphy, BSc, MD, FRCPC, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto General Hospital/ University Health Network, Toronto, Ontario, Canada